CLINICAL TRIAL: NCT03282708
Title: Comparative Study of Captive Great Ape and Human Intestinal Microbiomes
Brief Title: Comparative Study of Great Ape-caretaker Microbiome
Acronym: SHAPES-CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-081; ID-RCB: 2017-A00734-49 (Other: French national registration number of the study)
Record Dates: First submitted 2017-08-02; First posted 2017-09-14 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Human Intestinal Microbiome
Keywords: intestinal microbiome; captive great apes; human beings

STUDY DESIGN:
Intervention Model Description: 1 group of caretakers (9 volunteers). For this group: one sample collection of spontaneously produced fresh stools (of the approximate size of 3 green beans);
  1 group of caretakers (8 volunteers). For this group: no intervention (participant-observation only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiome (Experimental): Caretakers of captive great apes. One sample collection of spontaneously produced fresh stool (of an approximate size of 3 green beans).
  Data collection with self-administered questionnaire
  Interventions: Other: Fresh stool collection
- Anthropology (No Intervention): Caretakers of captive great apes. Two four-hour participant-observations of each caretaker's activities with captive great apes

INTERVENTIONS:
Other: Fresh stool collection — One sample collection of spontaneously produced fresh stool (of an approximate size of 3 green beans).
  Data collection with self-administered questionnaire
  Arms: Microbiome

SUMMARY:
The SHAPES-Captivity study seeks to identify metagenomic components of the intestinal microbiome shared by human beings and captive great apes living in proximity and in direct, daily contact. The investigators will determine the phylogenetic diversity of enterotypes (bacterial and viral) shared between human beings and great apes and will link these results with participant-observations of caretakers' activities (and contacts) with these great apes.

DETAILED DESCRIPTION:
The SHAPES-Captivity study seeks to identify metagenomic components of the intestinal microbiome shared by human beings and captive great apes living in proximity and in direct, daily contact. The SHAPES-Captivity is an extension of the SHAPES study (financed by the ANR in 2014), currently ongoing in central Africa (Democratic Republic of Congo, Cameroon, Gabon). In Cameroon, the investigators have collected stool samples from gorillas, chimpanzees and human beings using the same forest space so as to conduct an analysis of the overlap of their intestinal microbiome. The results of this analysis will be interpreted in light of anthropological and geographical evidence collected among people living in this region. SHAPES-Captivity will enable the investigators to use the same approach but this time, under conditions of great ape captivity. The investigators will thus obtain data concerning intestinal microbiome overlap between captive great apes and human caretakers working in a controlled environment and in daily, direct contact. The SHAPES-Captivity study will provide a positive control, which will eventually be compared to results from the SHAPES study. Although multiple studies have investigated the overlap between human-great ape intestinal microbiome (Moeller et al. 2012 ; Moeller et al. 2016), none of these studies have investigated people living in close proximity to great apes, either in a natural or captive setting. The investigators will determine the phylogenetic diversity of enterotypes (bacterial and viral) shared between human beings and great apes, and will link these results with their participant-observations of caretakers' activities (and contacts) with these great apes.

ELIGIBILITY:
Inclusion Criteria:

* For both Microbiome and Anthropology sub-study

  * Adult in good health
  * Currently working as a caretakers of captive great apes
* For Microbiome sub-study

  * Agree to autonomous collection of a stool sample
  * Agree to return the stool specimen inside of a designated, supplied postal container and box.
* For Anthropology sub-study:

  * Accept to be observed during his or her professional activity two times, each time for a duration of four hours by the researchers

Exclusion Criteria:

* For both Microbiome and Anthropology parts:

  * Protected adults, pregnant and nursing mothers will not be included.
* For Microbiome sub-study

  * Patients, especially those with gastrointestinal disorders (diarrhea), frequent and/or liquid stools, abdominal pain, nausea, vomiting, fever
  * Anyone diagnosed with a chronic disease
  * Anyone who has taken an antibiotic or antifungal treatment in the month preceding collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Microbiome comparison | Three years (September 2017-September 2020)
  The investigators will evaluate the components of the intestinal microbiome (viral and bacterial enterotypes) shared by human caretakers and captive great apes living in proximity on a daily basis. The percentage of overlap (of viral and bacterial families) between human subjects and great apes will be measured.

SECONDARY OUTCOMES:
Contact type investigation | Three years (September 2017-September 2020)
  The investigators will evaluate the type of physical contact between caretakers and great apes in captivity through participant-observations. This outcome will be measured through identified categories of physical contact.
Contact frequency investigation | Three years (September 2017-September 2020)
  The investigators will evaluate the frequency of physical contact between caretakers and great apes in captivity through participant-observations. This outcome will be measured by the number per category of physical contact.
Contact duration investigation | Three years (September 2017-September 2020)
  The investigators will evaluate the duration of physical contact between caretakers and great apes in captivity through participant-observations. This outcome will be measured by the duration (time) per individual contact.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Giles-Vernick, PhD, Study Director — Institut Pasteur
Locations (1):
- Institut Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No